CLINICAL TRIAL: NCT01249911
Title: Efficacy & Cost-Effectiveness of Lactobacillus Reuteri DSM 17938 Administration to Prevent the Risk of Respiratory or Gastrointestinal Infections in Child Day Care Centers: A Randomized, Double Blind, Placebo Control Trial (RDDCT).
Brief Title: Lactobacillus Reuteri DSM 17938 and Prevention of Respiratory and Gastrointestinal Infections in Mexican Infants
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Institute of Pediatrics, Mexico (Other Government)
Responsible Party: Pedro Gutierrez Castrellon, National Pediatric of Pediatrics, Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LreuteriMexico
Record Dates: First submitted 2010-11-28; First posted 2010-11-30 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Healthy Infants
Keywords: Infants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lreuteri (Experimental): Group of 130 infants allocated to receive L. reuteri DSM 17938 will be given at a dose of 5 drops containing 1x108 colony-forming units (CFU) once time per day in an oil formulation delivered from a drop bottle. In the active study product, freeze-dried L. reuteri is suspended in a mixture of pharmaceutical grade medium chain triglycerides and sunflower oil together with pharmaceutical grade silicon dioxide to give the product the correct rheological properties.
  Interventions: Dietary Supplement: Lreuteri
- Placebo (Placebo Comparator): The placebo consists of an identical formulation except that the L. reuteri is not present
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lreuteri — L. reuteri DSM 17938 will be given at a dose of 5 drops containing 1x108 colony-forming units (CFU) once time per day in an oil formulation delivered from a drop bottle. In the active study product, freeze-dried L. reuteri is suspended in a mixture of pharmaceutical grade medium chain triglycerides and sunflower oil together with pharmaceutical grade silicon dioxide to give the product the correct rheological properties.
  Arms: Lreuteri
Other: Placebo — The placebo consists of an identical formulation except that the L. reuteri is not present
  Arms: Placebo

SUMMARY:
Randomized, doble blind, clinical, controlled trial aimed to investigate the role of Lactobacillus reuteri DSM 17938 in the prevention of gastrointestinal and respiratory tract infections in mexican children who attend day care centers.

Primary Outcome: The primary outcome will be "days with diarrhoea". Secondary Outcomes: a) Days with respiratory tract infections (RTI); b) Days of absences from day care centre; c) Days of antibiotic use; d) Days of medical office visits or emergency visits; and e) Direct and Indirect costs.

Methods: Prospective, randomized, double blind, placebo controlled trial to realize in 260 healthy term infants, born at term (≥36 weeks of gestation), 6 to 36 months old, who will be recruit from Child Care Centers in Mexico and randomly allocated to receive either 1 x 108 colony-forming units of Lactobacillus reuteri DSM 17938 or placebo, each day for 12 weeks, follow up for other additionally 12 weeks of observation. Days with respiratory tract infections (RTI); days of absences from day care centre; days of antibiotic use; days of medical office visits or emergency visits; and direct and Indirect costs will be compare between groups using bi-variate, multiple lineal regression analysis and cost-effectiveness analysis

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants
* Born at term (≥36 weeks of gestation)
* Any gender
* 6 to 36 months old
* Same socioeconomic background
* Written informed consent from parents or legal guardians

Exclusion Criteria:

* Birth weight <2500 g
* Congenital anomalies
* Chronic diseases
* Failure to thrive
* Allergy or atopic disease
* Recent (within the preceding 4 weeks) exposure to probiotics, prebiotics, or antibiotics.
* Concurrent participation in other clinical trials

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 269 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-04 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
days with diarrhoea | January 2011 to June 2011
  Diarrhoea is defined as 3 or more loose or watery stools within 24 hours with or without vomiting. Days with diarrhoea is defined as the total amount of days with diarrhoea since the beginning of the study products administration until the last visit occurs. If liquid or loose stools is present a notification shall be made to the principal investigator.

SECONDARY OUTCOMES:
Days with respiratory tract infections (RTI) | January 2011 to June 2011
  Total amount of days with any RTI (common cold, rhinitis, acute rhinosinusitis, otitis, pharyngitis, tonsillitis, laryngitis, traqueítis, bronchiolitis, pneumonia), reported since the beginning of the study products administration until the last visit occurs
Days of absences from day care centre | January 2011 to June 2011
  Total amount of days of absences from the day care centre during the study, secondary to the presence of a gastrointestinal episode or RTI, reported since the beginning of the study products administration until the last visit occurs
Days of antibiotic use | January 2011 to June 2011
  Total amount of days of antibiotic use during the study, secondary to the presence of a gastrointestinal episode or RTI, reported since the beginning of the study products administration until the last visit occur
Days of medical office visits or emergency visits | January 2011 to June 2011
  Total amount of medical office visits or emergency visits during the study, secondary to the presence of a gastrointestinal episode or RTI, reported since the beginning of the study products administration until the last visit occurs.
Direct and Indirect costs | January 2011 to June 2011
  Total amount of money spent by hospital or parents (or guardians) during the study and secondary to the presence of a gastrointestinal episode or RTI, reported since the beginning of the study products administration until the last visit occur

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Gutierrez-Castrellon, MD, MSc, DSc, Principal Investigator — National Insitute of Pediatrics, Mexico; Gabriel Lopez Velazquez, PhD, Study Director — National Institute of Pediatrics, Mexico

REFERENCES:
- [Background] Savino F, Cordisco L, Tarasco V, Palumeri E, Calabrese R, Oggero R, Roos S, Matteuzzi D. Lactobacillus reuteri DSM 17938 in infantile colic: a randomized, double-blind, placebo-controlled trial. Pediatrics. 2010 Sep;126(3):e526-33. doi: 10.1542/peds.2010-0433. Epub 2010 Aug 16. PMID 20713478
- [Background] Coccorullo P, Strisciuglio C, Martinelli M, Miele E, Greco L, Staiano A. Lactobacillus reuteri (DSM 17938) in infants with functional chronic constipation: a double-blind, randomized, placebo-controlled study. J Pediatr. 2010 Oct;157(4):598-602. doi: 10.1016/j.jpeds.2010.04.066. Epub 2010 Jun 12. PMID 20542295
- [Background] Indrio F, Riezzo G, Raimondi F, Bisceglia M, Cavallo L, Francavilla R. Effects of probiotic and prebiotic on gastrointestinal motility in newborns. J Physiol Pharmacol. 2009 Dec;60 Suppl 6:27-31. PMID 20224148
- [Background] Abrahamsson TR, Sinkiewicz G, Jakobsson T, Fredrikson M, Bjorksten B. Probiotic lactobacilli in breast milk and infant stool in relation to oral intake during the first year of life. J Pediatr Gastroenterol Nutr. 2009 Sep;49(3):349-54. doi: 10.1097/MPG.0b013e31818f091b. PMID 19525871
- [Background] Bottcher MF, Abrahamsson TR, Fredriksson M, Jakobsson T, Bjorksten B. Low breast milk TGF-beta2 is induced by Lactobacillus reuteri supplementation and associates with reduced risk of sensitization during infancy. Pediatr Allergy Immunol. 2008 Sep;19(6):497-504. doi: 10.1111/j.1399-3038.2007.00687.x. Epub 2008 Jan 22. PMID 18221472
- [Background] Abrahamsson TR, Jakobsson T, Bottcher MF, Fredrikson M, Jenmalm MC, Bjorksten B, Oldaeus G. Probiotics in prevention of IgE-associated eczema: a double-blind, randomized, placebo-controlled trial. J Allergy Clin Immunol. 2007 May;119(5):1174-80. doi: 10.1016/j.jaci.2007.01.007. Epub 2007 Mar 8. PMID 17349686
- [Background] Savino F, Pelle E, Palumeri E, Oggero R, Miniero R. Lactobacillus reuteri (American Type Culture Collection Strain 55730) versus simethicone in the treatment of infantile colic: a prospective randomized study. Pediatrics. 2007 Jan;119(1):e124-30. doi: 10.1542/peds.2006-1222. PMID 17200238
- [Background] Weizman Z, Asli G, Alsheikh A. Effect of a probiotic infant formula on infections in child care centers: comparison of two probiotic agents. Pediatrics. 2005 Jan;115(1):5-9. doi: 10.1542/peds.2004-1815. PMID 15629974
- [Background] Rosenfeldt V, Benfeldt E, Valerius NH, Paerregaard A, Michaelsen KF. Effect of probiotics on gastrointestinal symptoms and small intestinal permeability in children with atopic dermatitis. J Pediatr. 2004 Nov;145(5):612-6. doi: 10.1016/j.jpeds.2004.06.068. PMID 15520759
- [Background] Fass RJ, Plouffe JF, Russell JA. Intravenous/oral ciprofloxacin versus ceftazidime in the treatment of serious infections. Am J Med. 1989 Nov 30;87(5A):164S-168S. doi: 10.1016/0002-9343(89)90050-8. PMID 2589361
- [Background] Rosenfeldt V, Michaelsen KF, Jakobsen M, Larsen CN, Moller PL, Tvede M, Weyrehter H, Valerius NH, Paerregaard A. Effect of probiotic Lactobacillus strains on acute diarrhea in a cohort of nonhospitalized children attending day-care centers. Pediatr Infect Dis J. 2002 May;21(5):417-9. doi: 10.1097/00006454-200205000-00013. PMID 12150179
- [Background] Rosenfeldt V, Michaelsen KF, Jakobsen M, Larsen CN, Moller PL, Pedersen P, Tvede M, Weyrehter H, Valerius NH, Paerregaard A. Effect of probiotic Lactobacillus strains in young children hospitalized with acute diarrhea. Pediatr Infect Dis J. 2002 May;21(5):411-6. doi: 10.1097/00006454-200205000-00012. PMID 12150178
- [Background] Shornikova AV, Casas IA, Mykkanen H, Salo E, Vesikari T. Bacteriotherapy with Lactobacillus reuteri in rotavirus gastroenteritis. Pediatr Infect Dis J. 1997 Dec;16(12):1103-7. doi: 10.1097/00006454-199712000-00002. PMID 9427453
- [Background] Shornikova AV, Casas IA, Isolauri E, Mykkanen H, Vesikari T. Lactobacillus reuteri as a therapeutic agent in acute diarrhea in young children. J Pediatr Gastroenterol Nutr. 1997 Apr;24(4):399-404. doi: 10.1097/00005176-199704000-00008. PMID 9144122
- [Derived] Gutierrez-Castrellon P, Lopez-Velazquez G, Diaz-Garcia L, Jimenez-Gutierrez C, Mancilla-Ramirez J, Estevez-Jimenez J, Parra M. Diarrhea in preschool children and Lactobacillus reuteri: a randomized controlled trial. Pediatrics. 2014 Apr;133(4):e904-9. doi: 10.1542/peds.2013-0652. Epub 2014 Mar 17. PMID 24639271